CLINICAL TRIAL: NCT00250783
Title: Pre-Clinical Models in Gynecological Tumors: A Tissue Repository
Brief Title: Pre-Clinical Models in Gynecological Tumors A Tissue Repository
Status: Completed | Type: Observational
Sponsor: University of New Mexico (Other)
Responsible Party: Sponsor
Other Study IDs: 2902C
Record Dates: First submitted 2005-11-04; First posted 2005-11-08 (Estimated); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Endometrial Neoplasms; Uterine Neoplasms
Keywords: Corpus Uteri; Endometrium; Cancer
MeSH Terms: conditions — Endometrial Neoplasms; Uterine Neoplasms; Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Tumor and normal tissues, ascites, and/or serum, and/or urine from women with malignant or premalignant gynecological conditions for which they are undergoing medically-indicated surgery, and normal tissues from women without malignancy who volunteer to donate serum and/or tissue at the time of medically indicated surgery
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to provide a repository for long-term storage of endometrial cancer tumor and normal tissue, ascites and serum. This material will be used in studies to better understand the molecular biology of endometrial cancer.

DETAILED DESCRIPTION:
BACKGROUND AND RATIONALE

This protocol will create a central repository for banking tumor and other tissues as well as serum from patients with uterine corpus tumors. In addition, this protocol will also serve as a central repository for serum and tissue to healthy post-menopausal and peri-menopausal controls.

There will be an "internal" bank. The internal bank will have samples available to UNM investigators.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing hysterectomy, or who have endometrial cancer, and are under routine surveillance.
* Patients may have received prior hormonal, cytotoxic chemotherapy, irradiation or surgical therapy.
* Healthy post-menopausal and peri-menopausal women.
* A consent form must be signed by the patient prior to study entry.

Exclusion Criteria:

Study Patients:

* Patients who do not have primary uterine corpus tumors.
* Patients with less than one gram of tumor tissue available to procurement.

Controls:

* Patients unwilling to have their medical records reviewed for height, weight, and general medical history (see attached data sheets).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: tumor and normal tissues, ascites, and/or serum, and/or urine from women with malignant or premalignant gynecological conditions for which they are undergoing medically-indicated surgery, and normal tissues from women without malignancy who volunteer to donate serum and/or tissue at the time of medically indicated surgery.
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2002-07 (Actual); Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Harriet Smith, MD, Principal Investigator — University of New Mexico
Locations (1):
- University of New Mexico, Albuquerque, New Mexico, United States